CLINICAL TRIAL: NCT05294198
Title: Beetroot Extract and Its Influence on Cardiovascular and Autonomic Recovery From the Effort in Healthy Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pernambuco (Other)
Responsible Party: Principal Investigator, Cicero Jonas R Benjamim, Nutritionist, University of Pernambuco
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: PX086
Record Dates: First submitted 2022-03-04; First posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Healthy Males

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Beet protocol (Experimental): Beta vulgaris L. extract (600mg)
  Interventions: Dietary Supplement: Beetroot extract
- Placebo protocol (Placebo Comparator): Starch (600mg)
  Interventions: Dietary Supplement: Beetroot extract

INTERVENTIONS:
Dietary Supplement: Beetroot extract — Beetroot extract capsule

SUMMARY:
There is no evidence that beetroot extract (Beta vulgaris L.) is advantageous for the recovery of cardiovascular parameters and the autonomic nervous system (ANS) after submaximal aerobic exercise. The objective of this study is to evaluate the effect of beetroot extract supplementation on the recovery of cardiorespiratory and autonomic parameters after a submaximal aerobic exercise session. Healthy male adults will perform a cross-over, randomized, double-blind, and placebo-controlled trial. Beetroot extract (600mg) or placebo (600mg) will be ingested 90 minutes before evaluation in randomized days. Systolic blood pressure (SBP), diastolic blood pressure (DBP), pulse pressure (PP), mean arterial pressure (MAP), heart rate (HR), and HR variability (HRV) indexes will be recorded at Rest and during 60 minutes of recovery from exercise.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males;
* Physically active according to International Physical Activity Questionnaire (IPAQ);
* 18 to 30 old years.

Exclusion Criteria:

* Body mass index BMI <18.5kg/m² and >29.9kg/m²;
* Smokers;
* Subjects undergoing pharmacotherapies;
* Musculoskeletal, metabolic, renal diseases;
* Root mean squared standard deviation of R-R intervals <15 milliseconds.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
Heart rate variability values (milliseconds) | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
Systolic and diastolic blood pressure values (mmHg) | Through study completion, an average of 1 year
Heart rate values (beats per minute) | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Cicero Benjamim, nutricionist, Principal Investigator — University of Pernambuco
Locations (1):
- University of Pernambuco, Petrolina, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: Undecided